CLINICAL TRIAL: NCT04124016
Title: Metabotypes in the Urinary Excretion of Flavan-3-ol Metabolites
Brief Title: Metabotypes in the Urinary Excretion of Flavan-3-ol Metabolites: "Metanols"
Acronym: Metanols
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Professor Furio Brighenti, Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 796/2018/SPER/UNIPR
Record Dates: First submitted 2019-09-03; First posted 2019-10-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Diet Modification
Keywords: flavan-3-ol; phenyl-y-valerolactones; catechins; metabotype; gas production; gut microbiota
MeSH Terms: interventions — Inulin; Tea; Grape Seed Extract

STUDY DESIGN:
Intervention Model Description: single-dose, partially randomized, cross over design with 4 consecutive treatments
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inulin (Experimental): Inulin_ extract of chicory fermentable fiber
  Interventions: Dietary Supplement: Inulin
- green tea extract (Experimental): green tea extract_rich in tri-hydroxylated flavan-3-ol monomers (1 mmol of PVL precursor)
  Interventions: Dietary Supplement: green tea extract
- grape seed (Experimental): grape seed extract - rich in di-hydroxylated flavan-3-ol monomers (1 mmol of PVL precursors)
  Interventions: Dietary Supplement: grape seed
- grape seed exctract (Experimental): grape seed extract - rich in di-hydroxylated flavan-3-ol oligomers (1 mmol of PVL precursors)
  Interventions: Dietary Supplement: grape seed extract

INTERVENTIONS:
Dietary Supplement: Inulin — Powder of inulin fractions dissolved into 250 ml of water
  Arms: Inulin
Dietary Supplement: green tea extract — Powder of green tea extract dissolved into 200 ml of water
  Arms: green tea extract
Dietary Supplement: grape seed — Powder of grape seed extract (rich in di-hydroxylated flavan-3-ol monomers) dissolved into 200 ml of water
  Arms: grape seed
Dietary Supplement: grape seed extract — Powder of grape seed extract (rich in di-hydroxylated flavan-3-ol oligomers) dissolved into 200 ml of water
  Arms: grape seed exctract

SUMMARY:
Flavan-3-ols are the main source of flavonoids in Western diets. They are characteristic compounds of tea, cocoa, wine, apple, pears, etc. In plant-based foods, they occur as simple monomers or as oligomers and polymers of up to 50 units (also known as proanthocyanidins or condensed tannins). When ingested, both monomeric and high molecular weight flavan-3-ols are poorly absorbed and metabolized in the first gastrointestinal tract, reaching the colon and becoming a suitable substrate for the local microbiota. These compounds undergo an extensive microbial metabolism leading to the formation of hydroxyphenyl-γ- valerolactones (PVLs), which are then absorbed by colonocytes before reaching the liver and being converted into phase II conjugated metabolites. Since the microbiota composition varies among individuals, it results in differences in the production of PVLs and, consequently, the health effects of flavan-3-ols might change at an individual level.

Another factor of variability might be due to a different asset in the fermentation of indigestible dietary carbohydrates, which are known to modify colonic pH through the production of short-chain fatty acids and may result in different profiles of gas production (i.e. hydrogen and methane), possibly affecting the bioconversion of flavan-3-ols as well. Nevertheless, these multiple variabilities are poorly understood to date.

DETAILED DESCRIPTION:
The study will be a single-dose, partially randomized, cross-over design, with 4 consecutive treatments. The study includes 4 phases where each volunteer will consume a specific dose of one of the products chosen for the study. Each volunteer will consume each product once, for a total of 4 different occasions. The products will be a food extract consisting of chicory fermentable fiber (inulin) fractions followed by three food extracts rich in a different type of flavan-3-ols, consumed at three different occasions and in random order.

Volunteers will be asked to provide once a fecal sample, taken from the first daily defecation, which will be analyzed for fecal microbiota composition. They will also undergo a Breath gases day profile in order to evaluate the effect of inulin consumption on colonic fermentation and breath-gases production. These two analyses (fecal samples microbial composition and breath-gases production) will serve to characterize the volunteers' gut microbiota composition and functionality. In detail, during the 48-h before the fecal and breath samples collections, volunteers will be asked to avoid a high level of fiber and (poly)phenols (to facilitate adherence to the dietary restrictions, a list of permitted and forbidden foods will be supplied. To check dietary compliance, a 2- days dietary record of the 2 days prior to each sampling day will be used.

The morning of the first treatment, volunteers will arrive, after an overnight fast, and they will deliver the fresh fecal sample. After that, one sample of forced end-expiratory samples of alveolar air will be collected. Then, they will be given a standardized test breakfast consisting of 12 g of food extract of chicory inulin fractions dissolved into 250 g water and a fermentable fiber-free, (poly)phenol-free, nutritionally-balanced solid meal. They will be asked to consume the entire breakfast within 15 minutes. At hourly intervals for 11 hours after breakfast, forced end-expiratory samples of alveolar air will be collected. During the whole test, all subjects will refrain from smoking, sleeping, exercising and eating foods or meals other than the ones provided by the staff. Five hours after starting the test, volunteers will eat a fermentable fiber-free nutritionally-balanced standardized lunch provided by the study staff.

Subsequently, on three distinct occasions and with one-week wash-out between different treatments, each participant will randomly consume a dose of flavan-3-ol rich extracts. Each test day, participants, after fasting baseline urine collection, will receive the dose of one of the food extract rich in flavan-3-ols (1 mmol of PVL precursors) dissolved into 200 mL of water. Then, the same standardized breakfast (pre-packaged (poly)phenol-free snack) will be provided to subjects. After breakfast, volunteers will be allowed to leave and to perform the successive urine collections on their own. Urine samples will be collected at selected intervals of time along the 24 h following the extract ingestion. In addition, urine sampling will continue in a subgroup of volunteers for the successive 24 h to evaluate the evolution of metabotypes from 24 to 48h. This subgroup will be composed of the first 30 participants enrolled in the study.

Subjects will be asked to follow a (poly)phenol-poor diet 48-h before each test day and while sampling (to facilitate adherence to the dietary restrictions, a list of permitted and forbidden foods will be supplied; to check dietary compliance, a 3/4-days dietary record of the 2 days prior to each sampling day and of the sampling day(s), depending on the subgroup the subject belongs to, will be used.

At the end of all treatments, and on the basis of the results of gas samples analysis, one subgroup of methane producer volunteers (number=5) and one of non-methane producers (numnber=5) will be asked to provide one further faecal sample, taken from the first daily defecation for In Vitro analysis of short-chain fatty acids and gas production after incubation with different mixes of Inulin and Polyphenols used during the In Vivo part of the study . Volunteers will be asked to follow a diet poor in (poly)phenols and fermentable fiber for 2 days before fecal donation.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Both genders
* Healthy
* BMI > 18.5
* BMI < 30

Exclusion Criteria:

* Metabolic disorder or surgeries of liver, kidney or gastrointestinal tract
* Immunodeficiency
* Food intolerance or allergies
* Regular consumption of medication
* Antibiotic therapy within the last 3 months
* Use of food supplements, including pro- and prebiotics
* Intense physical activity (PAL ≥ 2.10)
* Pregnancy
* Lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-12-27 (Estimated)

PRIMARY OUTCOMES:
Assessing the formation of urinary metabotypes of flavan-3-ol colonic metabolites | AUC for 24 hours (sum of 0-180; 180-360; 360-540; 540-720; 720-1440 minutes)
  Assessing the variability of the area under the curve of the urinary concentration of some phenolic metabolites ( tri- and di-hydroxyphenyl-γ-valerolactones and 3-hydroxyphenylpropionic acids (umol)) after consumption of 3 different sources of flavan-3-ols by using data-driven clustering.

SECONDARY OUTCOMES:
Evolution over the time of the metabolites of flavan-3-ols in urine samples | AUC for 48 hours (sum of 0-180; 180-360; 360-540; 540-720; 720-1440; 1440-2160; 2160-2880; 2880 minutes)
  Assessed by using UHPLC-MSn for individual detection and quantification.
Identification of Firmicutes, bacteroidetes and Archea in faecal samples of participants | Baseline
  Firmicutes, Bacteroidetes and Archea main species assessed by an optimized 16S rRNA gene-based analysis protocol.
Evaluation of inter-individual differences on breath-gases production (hydrogen and methane) on alveolar air samples | AUC for 12 hours; (sum of 60; 120; 180; 240; 300; 360; 420; 480; 540; 600; 660; 720 minutes)
  Performed by using a hydrogen/methane analyser
Correlations between colonic fermentation, gas production and microbiota composition and metabotypes | 24 hours
  multiple correlation between in vitro short chain fatty acids and gas production, microbiota composition and metabotype through PCA and PLS-DA.
In vitro variation of gases production by fermentable dietary fibre in presence of polyphenols using faecal starters | Baseline
  Gasses production will be assessed using a hydrogen/methane analyser
In vitro variation of short chain fatty acids production of fermentable dietary fibre in presence of polyphenols using faecal starters | Baseline
  Short chains fatty acids will be quantified using GC-MS
Untargeted metabolomics on urine samples | 24 hours
  Metabolomics will be carried out in urine using HR-LC-MS/MS to unravel the potential metabolic pathways of molecules present after the consumption of the different sources of flavan-3-ols.

CONTACTS AND LOCATIONS:
Overall Officials: Furio FB Brighenti, Professor, Principal Investigator — University of Parma; Daniele DR Del Rio, Professor, Study Director — University of Parma; Pedro Miguel PM Mena Parreño, Ph.D., Study Director — University of Parma; Rossella RD Dodi, M. Sc., Study Director — University of Parma
Locations (1):
- University of Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: Undecided